CLINICAL TRIAL: NCT03372993
Title: A Post-Marketing, Observational Study in Iran to Determine the Immunogenicity Status in Patients Who Have Received rFVIIa AryoSeven.
Brief Title: Prospective, Non-interventional Study to Evaluate Immunogenicity of AryoSeven
Status: Completed | Type: Observational
Sponsor: AryoGen Pharmed Co. (Industry)
Responsible Party: Sponsor
Other Study IDs: ARY2016-01
Record Dates: First submitted 2017-12-05; First posted 2017-12-14 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2020-07

CONDITIONS: Hemophilia A With Inhibitor; Hemophilia B With Inhibitor; Factor VII Deficiency; Glanzmann's Thrombasthenia
MeSH Terms: conditions — Factor VII Deficiency; Thrombasthenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma for PT based Bethesda assay.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the immunogenicity of the biosimilar rFVIIa (AryoSeven) in subjects receiving AryoSeven in real-life clinical practice.

DETAILED DESCRIPTION:
This is a Non-interventional, observational, prospective evaluation of immunogenicity (neutralizing antibodies toward FVII) of patients with Hemophilia A or B with inhibitors, Factor VII Deficiency, Glanzmann's thrombasthenia, who have received one or more dose of AryoSeven in the daily practice. This study is conducted in Iran where AryoSeven is available on the market since 21-8-2012 and NovoSeven is no longer available since 2013. Patients will be retrieved from the Iranian Registry of Hemophilia patients of MATHA (Iranian Hemophilia and Thrombophilia Association, Tehran, Iran). The Registry Patient Screener will sequentially review patients in the Registry to identify patients who have received treatment with AryoSeven, in reverse chronological order of inclusion in the registry, starting from a date 6 months prior to the date of this study and until when the sample size to enroll (200 patients) is completed.

Patients identified will be called for a visit (Screening visit) for providing informed consent, interview, and blood sampling collection for prospective immunogenicity testing. Retrospective data collection, including previous immunogenicity status and the number of exposure days, will be performed on hospital records, patient diary. Immunogenicity will be tested by a centralized laboratory in Iran using the PT-based Bethesda assay.

Patients will be enrolled if they had an immunogenicity test negative, performed at the earliest time after NovoSeven was no longer available in Iran. Patients who do not have a previous negative immunogenicity test will be enrolled if negative at immunogenicity test performed during screening for this study.

Patients enrolled will be followed for at least 12 months for immunogenicity and Adverse Drug Reactions.

Patients who have a positive previous immunogenicity test or results positive at immunogenicity test performed at Screening (patients without a previous immunogenicity test), will not be enrolled, but registered and followed for 12 months (or longer) to collect data on the natural history of their disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Hemophilia A or B with inhibitors, Factor VII Deficiency, Glanzmann's thrombasthenia
* Treated with AryoSeven in the daily practice,
* Signed informed consent (parents for children).
* an immunogenicity test negative, performed at the earliest time after NovoSeven was no longer available in Iran. Patients who do not have a previous negative immunogenicity test should be enrolled if negative at immunogenicity test performed during screening for this study.

Exclusion Criteria:

* Patients who received NovoSeven for any indication at any time before inclusion in the study, until an immunogenicity test excluded the development of immunogenicity related to NovoSeven.
* Parallel participation in another experimental drug trial.
* Parallel participation in another marketed drug trial (except for AryoSeven) that may affect the immunogenicity endpoint of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Hemophilia A or B with inhibitors, Factor VII Deficiency, Glanzmann's thrombasthenia, who have received one or more dose of AryoSeven in the daily practice and are negative at immunogenicity testing (antibodies neutralizing FVII).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Immunogenicity (neutralising antibodies toward FVII) | On plasma samples obtained 12 months after patient inclusion.
  Immunogenicity will be assessed with the PT based Bethesda assay. In case of positive results, an inhibitor retesting using a second separately drawn sample as confirmatory measurement will be performed by a different specialised laboratory.

SECONDARY OUTCOMES:
Adverse Drug Reactions | Adverse Drug Reactions will be monitored throughout the trial, from patient inclusion up to 12 months follow-up.
  Adverse Drug Reactions related to the administration of AryoSeven reported by patients.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Faranoush, MD, Study Director — Hazrat Rasool Akram Hospital, MAHAK Children's Hospital, Iran University of Medical Sciences, Tehran
Locations (2):
- Iran (2):
  - Iranian Blood Transfusion Organization (IBTO), Tehran
  - MAHTA (Iranian Hemophilia and Thrombophilia Association), Tehran